CLINICAL TRIAL: NCT05978726
Title: Ticagrelor Versus Clopidogrel for Coronary Microvascular Dysfunction in Patients With Acute Myocardial Infarction: A Retrospective Study Based on the Angiography-derived Index of Microcirculatory Resistance
Brief Title: Ticagrelor Versus Clopidogrel for CMD in Patients With AMI: A Retrospective Study Based on the Angio-IMR
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2023007
Record Dates: First submitted 2023-07-31; First posted 2023-08-07 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-07

CONDITIONS: Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease | interventions — Aspirin; Clopidogrel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- ticagrelor maintenance treatment group: Patients received dual antiplatelet therapy (DAPT) with aspirin 100mg daily and ticagrelor 90mg twice daily for at least 9 months after PCI. Angio-IMR assessment was performed after primary PCI and during routine follow-up coronary angiography.
  Interventions: Drug: Dual antiplatelet therapy with aspirin and either ticagrelor or clopidogrel
- clopidogrel maintenance treatment group: Patients received dual antiplatelet therapy (DAPT) with aspirin 100mg daily and clopidogrel 75mg once daily for at least 9 months after PCI. Angio-IMR assessment was performed after primary PCI and during routine follow-up coronary angiography.

INTERVENTIONS:
Drug: Dual antiplatelet therapy with aspirin and either ticagrelor or clopidogrel — Patients with acute myocardial infarction randomly received dual antiplatelet therapy with with aspirin 100mg daily and either ticagrelor 90mg twice daily or clopidogrel 75mg once daily for at least 9 months after PCI as needed.
  Groups: ticagrelor maintenance treatment group

SUMMARY:
Coronary microvascular dysfunction (CMD) is increasingly recognized as an important indicator for long-term prognosis in patients with acute myocardial infarction (AMI). The angiography-derived index of microcirculatory resistance (angio-IMR) is a novel guidewire-free measure for CMD in patients with AMI. Ticagrelor has recently been suggested to have additional benefits on coronary microcirculation beyond its antiplatelet effect. This study was designed to compare the protective effects of ticagrelor and clopidogrel on CMD and prognostic impact in patients with AMI, using the angio-IMR as a novel assessment tool.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were diagnosed with AMI, including STEMI and NSTEMI, and underwent successful PCI and routine follow-up coronary angiography at the Second Affiliated Hospital of Zhejiang University School of Medicine between June 1, 2017 and May 31, 2020.

Exclusion Criteria:

* 1) prior treatment with any P2Y12 inhibitor;
* 2) need for long-term oral anticoagulation therapy;
* 3) previous coronary artery bypass grafting (CABG);
* 4) chronic renal dysfunction with estimated glomerular filtration rate (eGFR) <30 mL/ (min·1.73 m2) or on hemodialysis;
* 5) liver cirrhosis ≥Child-Pugh B class;
* 6) cancer;
* 7) adjustment of dual antiplatelet therapy (DAPT) during follow-up;
* 8) inadequate coronary angiographic images.

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: We retrospectively enrolled patients who were diagnosed with AMI, including STEMI and NSTEMI, and underwent successful PCI and routine follow-up coronary angiography at the Second Affiliated Hospital of Zhejiang University School of Medicine between June 1, 2017 and May 31, 2020. The diagnosis of AMI was based on current clinical guidelines. All patients were pretreated with oral aspirin 300mg and a loading dose of ticagrelor 180mg or clopidogrel 300mg before PCI. Patients received dual antiplatelet therapy (DAPT) with aspirin 100mg daily and either ticagrelor 90mg twice daily or clopidogrel 75mg once daily for at least 9 months after PCI. Patients were divided into clopidogrel group and ticagrelor group according to the post-PCI antiplatelet maintenance therapy.
Sampling Method: Non-Probability Sample
Enrollment: 325 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
The improvement of angio-IMR | within 24 months post-PCI
  Difference between Angio-IMR at follow-up coronary angiography and Angio-IMR after PCI

SECONDARY OUTCOMES:
Readmission for heart failure | Within 24 months post-PCI
  Readmission for an acute exacerbation of chronic heart failure or acute heart failure
Myocardial reinfarction | Within 24 months post-PCI
  Another myocardial infarction with elevated myocardial enzymes and abnormal electrocardiograms
Target vessel revascularization | Within 24 months post-PCI
  Repeat revascularization was performed because of ischemia in the target-vessel territory
Non-target vessel revascularization | Within 24 months post-PCI
  Repeat revascularization was performed because of ischemia in the non-target vessel territory
Cerebral hemorrhage | Within 24 months post-PCI
  The occurrence of cerebral hemorrhage during the follow-up period was based on imaging CT and MRI
Other bleeding events | Within 24 months post-PCI
  Bleeding events such as gingival bleeding, skin bleeding, and gastrointestinal bleeding and so on, occurred during the follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Jun Jiang, MD, PhD, Study Director — Second affiliated Hospital Zhejiang University School of Medicine
Locations (1):
- Second affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jiang J, Li C, Hu Y, Li C, He J, Leng X, Xiang J, Ge J, Wang J. A novel CFD-based computed index of microcirculatory resistance (IMR) derived from coronary angiography to assess coronary microcirculation. Comput Methods Programs Biomed. 2022 Jun;221:106897. doi: 10.1016/j.cmpb.2022.106897. Epub 2022 May 18. PMID 35636354
- [Background] Choi KH, Dai N, Li Y, Kim J, Shin D, Lee SH, Joh HS, Kim HK, Jeon KH, Ha SJ, Kim SM, Jang MJ, Park TK, Yang JH, Song YB, Hahn JY, Doh JH, Shin ES, Choi SH, Gwon HC, Lee JM. Functional Coronary Angiography-Derived Index of Microcirculatory Resistance in Patients With ST-Segment Elevation Myocardial Infarction. JACC Cardiovasc Interv. 2021 Aug 9;14(15):1670-1684. doi: 10.1016/j.jcin.2021.05.027. PMID 34353599
- [Derived] Fang J, Zhang Y, Zheng Y, Chen D, Yidilisi A, Ji R, Xiang J, Zhang X, Jiang J. Comparison of Ticagrelor with Clopidogrel on Coronary Microvascular Dysfunction Following Acute Myocardial Infarction Using Angiography-Derived Index of Microcirculatory Resistance. Cardiovasc Drugs Ther. 2025 Oct;39(5):1097-1111. doi: 10.1007/s10557-024-07619-4. Epub 2024 Sep 2. PMID 39222277